CLINICAL TRIAL: NCT02347904
Title: Feasibility Study of Adjuvant Treatment With S-1 and Oxaliplatin in Patients With Resectable Esophageal Cancer
Acronym: SOX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, H.W.M. van Laarhoven, Prof. Dr. H.W.M. van Laarhoven, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL49889.018.14
Record Dates: First submitted 2014-12-16; First posted 2015-01-28 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer; Adjuvant treatment; S-1; Oxaliplatin; Feasibility
MeSH Terms: conditions — Esophageal Neoplasms | interventions — S 1 (combination); Oxaliplatin; tegafur-gimeracil-oteracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adjuvant S-1 and Oxaliplatin (Experimental): Adjuvant treatment with s-1 and oxaliplatin after neoadjuvant chemoradiation and esophagectomy in patients with resectable esophageal cancer
  Interventions: Drug: S-1 and Oxaliplatin

INTERVENTIONS:
Drug: S-1 and Oxaliplatin — Six courses of oxaliplatin (130 mg/m2) intravenously on day 1 and S-1 (25 mg/m2 b.i.d.) orally from day 1 to 14 every 3 weeks, starting within 12 weeks after esophagectomy
  Other Names: Teysuno

SUMMARY:
In this prospective single arm study the investigators will assess the feasibility of S-1 and Oxaliplatin as adjuvant treatment in patients with esophageal cancer.

The primary objective is to assess the feasibility of administering adjuvant S-1 and Oxaliplatin (SOX) in patients with esophageal cancer after neoadjuvant chemoradiotherapy with paclitaxel and carboplatin and esophagectomy. Primary end point is the percentage of patients completing the preplanned number of 6 cycles of SOX.

DETAILED DESCRIPTION:
Since the outcome of patients with esophageal cancer treated with neoadjuvant chemoradiation and surgery is still poor, strategies to improve survival should be explored. The benefit of adjuvant chemotherapy after neoadjuvant chemoradiotherapy followed by surgery is unknown. Preferably, such adjuvant chemotherapy regimen should consist of a non-cross resistant, well-tolerated schedule. For this purpose, the combination of S-1, an oral fluoropyrimidine, with oxaliplatin, may be of benefit, as each of these compounds have shown efficacy in gastroesophageal cancer. Also, importantly, the combination of S-1 with oxaliplatin (SOX) in advanced gastric cancer was well-tolerated. Nevertheless, it should be acknowledged that after major surgery for esophageal cancer, adjuvant treatment with combination chemotherapy may be hard to accomplish as was shown in the MAGIC trial for gastric cancer where less than half of all patients completed adjuvant therapy.

Therefore the investigators want to assess the feasibility of an adjuvant treatment scheme with S-1 and Oxaliplatin. When the proposed treatment scheme is feasible the potential benefit on survival will be evaluated in further studies. Feasibility is defined ≥50% of patients completing the pre-planned number of cycles

Study Objectives Primary Objective To assess the feasibility of administering adjuvant SOX in patients with esophageal cancer after neoadjuvant chemoradiotherapy with paclitaxel and carboplatin and esophagectomy

Secondary Objectives

1. Percentage of patients completing 6 cycles of S-1 (with or without oxaliplatin).
2. Dose modifications (ie, delays, dose reductions, or interruptions) for S-1.
3. Dose modifications (ie, delays, dose reductions, or interruptions) for oxaliplatin.
4. Dose intensity of S-1.
5. Dose intensity of oxaliplatin.
6. Toxicity.
7. Disease free survival.

Exploratory Objectives

1. Assessment of pharmacokinetics of S1 as predictive factors for efficacy and toxicity.
2. Potential biomarker development based on assessment of archived tumor tissue and blood samples and the proposed mechanism of action of study drugs.

ELIGIBILITY:
Inclusion Criteria:

* Radically resected adenocarcinoma of the esophagus
* Completed neoadjuvant treatment with paclitaxel 50 mg/m2 and carboplatin Area Under Curve (AUC) = 2 on days 1, 8, 15, 22 and 29 and radiotherapy to a total dose of 41.4 Gy in 23 fractions of 1.8 Gy, 5 fractions per week.
* Age ≥ 18 years
* WHO performance status 0-1
* Adequate bone marrow function (Hb ≥ 6.0 mmol/L, absolute neutrophil count ≥1.0 x 109/L, - platelets ≥ 100 x 109/L), renal function (serum creatinine ≤ 1.5x ULN and creatinine clearance, Cockroft formula, ≥30 ml/min), liver function (serum bilirubin ≤ 2 x Upper Limit Normal (ULN), serum transaminases ≤ 3 x).
* Negative pregnancy test in women with childbearing potential.
* Expected adequacy of follow-up.
* Written informed consent.

Exclusion Criteria:

* Any history or clinical signs of metastasis
* History of a second malignancy <5 years with the exception of adequately treated carcinoma of cervix or basal/squamous cell carcinoma of skin.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency or treatment within 4 weeks with DPD inhibitors, including sorivudine or its chemically related analogues such as brivudine.
* Significant cardiovascular disease < 1 yr before start of the study (symptomatic congestive heart failure, myocardial ischemia or infarction, unstable angina pectoris, serious uncontrolled cardiac arrhythmia, arterial thrombosis, cerebrovascular event, pulmonary embolism).
* Chronic active infection.
* Any other concurrent severe or uncontrolled disease preventing the safe administration of study drugs.
* Any impairment of gastrointestinal function or -disease that may significantly impair the absorption of oral drugs (i.e. uncontrolled nausea, vomiting, diarrhoea (defined as CTC grade 2 or higher), malabsorption syndrome, bowel obstruction, or inability to swallow tablets).
* Concomitant treatments: concomitant (or within 4 weeks before start of the study) administration of any other experimental drug under investigation; concurrent treatment with any other anti-cancer therapy.
* Continuous use of systemic immunosuppressive agents (except the use of corticosteroids as anti-emetic prophylaxis/treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
The percentage of patients completing the preplanned number of 6 cycles of SOX. | 24 months

SECONDARY OUTCOMES:
Percentage of patients completing 6 cycles of S-1 (with or without oxaliplatin) | 24 months
Dose modifications for S-1 | 24 months
  in terms of delay of treatment in weeks
Dose modifications for S-1 | 24 months
  in terms of dose reduction in percentage of orginal dose
Dose modifications for S-1 | 24 months
  in terms of number of interruptions of treatment
Dose modifications for Oxaliplatin | 24 months
  in terms of delay of treatment in weeks
Dose modifications for Oxaliplatin | 24 months
  in terms of dose reduction in percentage of orginal dose
Dose modifications for Oxaliplatin | 24 months
  in terms of number of interruptions of treatment
Dose intensity for S-1 | 24 months
  total received dose of S-1 in mg/m2 per week
Dose intensity for Oxaliplatin | 24 months
  total received dose of oxaliplatin in mg/m2 per week
Toxicity | 24 months
  in terms of CTCAE v4.0 criteria
Disease free survival | 24 months
  in months
Overall survival | 24 months
  in months

OTHER OUTCOMES:
AUC of S-1 | 24 months
  assessment of pharmacokinetics (Cmax/T1/2) in relation to toxicity in terms of CTCAE criteria and efficacy in terms of disease free survival

CONTACTS AND LOCATIONS:
Overall Officials: H WM van Laarhoven, MD,PHD,PHD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Medical Oncology, Amsterdam, Netherlands